CLINICAL TRIAL: NCT07242105
Title: Optimized Methods for Measuring Brain Excitability in Depression
Brief Title: Optimizing Brain Excitability in Depression
Acronym: TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Corey Keller, Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 72673-1; 1R01MH139650 (NIH)
Record Dates: First submitted 2025-11-11; First posted 2025-11-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: tms; eeg
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active TMS, Sham TMS with iEEG (Experimental): Neurosurgical participants receive both active single-pulse Transcranial Magnetic Stimulation (TMS) and sham single-pulse TMS delivered to predefined dlPFC sites while undergoing intracranial EEG recording. The order of active and sham stimulation is randomized.
  Interventions: Device: Active Single-Pulse TMS; Device: Sham Single-Pulse TMS; Other: Intracranial EEG (iEEG) Recording
- Sham TMS, Active TMS with iEEG (Experimental): Neurosurgical participants receive sham single-pulse TMS followed by active single-pulse TMS at predefined dlPFC sites during intracranial EEG recording. The order of stimulation conditions is randomized.
  Interventions: Device: Active Single-Pulse TMS; Device: Sham Single-Pulse TMS; Other: Intracranial EEG (iEEG) Recording
- Optimized TMS, Non-optimized TMS with EEG (Experimental): Participants receive both TARGET optimized single-pulse TMS and non-optimized (open-loop) single-pulse TMS to the dlPFC while undergoing concurrent scalp EEG. The sequence of optimized and non-optimized stimulation is randomized.
  Interventions: Device: TARGET-optimized TMS; Device: Non-optimized (Open-Loop) TMS; Other: EEG Recording
- Non-optimized TMS, Optimized TMS with EEG (Experimental): Participants receive non-optimized (open-loop) single-pulse TMS followed by TARGET optimized single-pulse TMS to the dlPFC with concurrent scalp EEG. The order of stimulation conditions is randomized.
  Interventions: Device: TARGET-optimized TMS; Device: Non-optimized (Open-Loop) TMS; Other: EEG Recording

INTERVENTIONS:
Device: Active Single-Pulse TMS — Single-pulse transcranial magnetic stimulation is delivered to the left dorsolateral prefrontal cortex using a MagVenture X100 stimulator and B65 A/P coil across predefined locations, coil angles, and stimulation intensities.
  Arms: Active TMS, Sham TMS with iEEG; Sham TMS, Active TMS with iEEG
Device: Sham Single-Pulse TMS — Sham single-pulse TMS is delivered using a flipped coil and concurrent scalp electrical stimulation to mimic auditory and somatosensory sensations without producing cortical stimulation.
  Arms: Active TMS, Sham TMS with iEEG; Sham TMS, Active TMS with iEEG
Device: TARGET-optimized TMS — Single-pulse TMS parameters (location, angle, and intensity) are adjusted in real time using the TARGET closed-loop algorithm based on concurrent EEG measurements to deliver optimized stimulation.
  Arms: Non-optimized TMS, Optimized TMS with EEG; Optimized TMS, Non-optimized TMS with EEG
Device: Non-optimized (Open-Loop) TMS — Single-pulse TMS is delivered using a predefined open-loop set of stimulation parameter combinations across multiple dlPFC locations, coil angles, and intensities without real-time adjustment.
  Arms: Non-optimized TMS, Optimized TMS with EEG; Optimized TMS, Non-optimized TMS with EEG
Other: EEG Recording — Participants undergo concurrent 64-channel TMS-compatible scalp EEG recording during stimulation to measure TMS-evoked neural responses.
  Arms: Non-optimized TMS, Optimized TMS with EEG; Optimized TMS, Non-optimized TMS with EEG
Other: Intracranial EEG (iEEG) Recording — Neurosurgical participants undergo intracranial EEG recording using clinically implanted electrodes during TMS to measure local and downstream neural activity.
  Arms: Active TMS, Sham TMS with iEEG; Sham TMS, Active TMS with iEEG

SUMMARY:
The goal of this study is to improve depression treatment by establishing reliable prefrontal excitability markers through Targeting with Automated Real-time Guidance for Enhancing TEPs (TARGET).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 65
* Diagnosis of major depressive disorder, assessed through a Structured Clinical Interview for DSM-5 (SCID-5)
* In a current depressive episode, assessed through a Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (SCID-5)
* Moderate-to-severe depression as indicated by a score between 11-20 on the Quick Inventory of Depressive Symptoms (QIDS)
* Must comprehend English well to ensure adequate comprehension of the EEG and TMS instructions, and of clinical scales
* No current or history of neurological disorders
* No seizure disorder or risk of seizures
* Neurosurgical patients: Men and women ages 18-65 with medication-refractory epilepsy who are admitted for phase II intracranial monitoring to detect a seizure focus will be considered appropriate for this study. Participants must have the intellectual capacity to understand the consent process and agree to the study.

Exclusion Criteria:

* Those with a contraindication for MRIs (e.g. implanted metal)
* History of head trauma with loss of consciousness
* History of seizures or on medications that reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium)
* Neurological or uncontrolled medical disease
* Any unstable medical condition
* Active substance abuse
* Diagnosis of psychotic or bipolar disorder
* A prior history of Electroconvulsive Therapy (ECT) failure
* History of suicide attempt in the past year
* Currently pregnant or breastfeeding
* Repetitive Transcranial Magnetic Stimulation (rTMS) treatment in the past six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Anterior EL-TEP Amplitude after single-pulse TMS (spTMS) | Baseline, end of spTMS (6 hours)
  Changes in Early Local TMS-Evoked Potentials (EL-TEP) following 6 hours of either active or sham spTMS between optimized and non-optimized stimulation conditions in the anterior dlPFC.
Changes in Posterior EL-TEP Amplitude after spTMS | Baseline, end of spTMS (6 hours)
  Changes in Early Local TMS-Evoked Potentials (EL-TEP) following 6 hours of either active or sham spTMS between optimized and non-optimized stimulation conditions in the posterior dlPFC.
Changes in intracranial TMS-Evoked Potential (iTEP) Amplitude after TMS-iEEG | Baseline, end of spTMS (20 minutes)
  Changes in the interaction between gyral/sulcal targets and coil angles (45 vs 90 degrees) on local dlPFC iTEP amplitude.

CONTACTS AND LOCATIONS:
Overall Officials: Corey J Keller, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No